CLINICAL TRIAL: NCT01809600
Title: Rituximab-Containing Immunochemotherapy for Burkitt's Lymphoma (BL) and High-Grade B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and BL
Brief Title: Retrospective Analysis of Rituximab-containing Immunochemotherapy for Burkitt's or Burkitt-like Lymphoma in Adults
Acronym: RBL
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Junshik Hong, Assistant Professor, Department of Internal Medicine, Gachon University Gil Medical Center
Other Study IDs: CISL-1203
Record Dates: First submitted 2013-03-08; First posted 2013-03-13 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Burkitt's Lymphoma; High-grade B-cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Burkitt's Lymphoma: should be diagnosed pathologically by WHO 2008 criteria
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study)

SUMMARY:
This retrospective study is aimed at evaluating the safety and efficacy of rituximab-containing immunochemotherapy in adult patients with Burkitt's lymphoma (BL) or high-grade B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and BL.

DETAILED DESCRIPTION:
Inclusion criteria

1. pathologically confirmed BL or BL-U by World Health Organization 2008 criteria
2. age >20 yrs
3. received rituximab+chemotherapy as first-line treatment
4. with measurable or evaluable lesion
5. with complete set of clinical and laboratory data for the analysis

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed Burkitt's lymphoma (BL) or High grade B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and BL (BL-U) by WHO 2008 criteria
2. age >20 yrs
3. received rituximab+chemotherapy as first-line treatment
4. with measurable or evaluable lesion

Exclusion Criteria:

1. patients with BL or BL-U previously treated with rituximab

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were treated with Burkitt's or Burkitt-like high-grade B-cell lymphoma in Republic of Korea
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Event-free survival | one year
  Event-free survival is measured from the time from treatment initiation to any treatment failure including disease progression, or discontinuation of treatment for any reason (eg, disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death)

SECONDARY OUTCOMES:
complete response rate | 1-year
  treatment response will be evaluated according to the Revised criteria for malignant lymphoma (Journal of Clinical Oncology 25:579-586)
overall survival | 1-year
  Overall survival is defined as the time from treatment initiation until death as a result of any cause
Grade 4 hematologic toxicities | one year
  toxicities will be graded according to Common Toxicity Criteria for Adverse Events (CTCAE) V.4.0. Hematologic toxicities planned to evaluated were; anemia (by hemoglobin), absolute neutrophil count, and platelet count

CONTACTS AND LOCATIONS:
Overall Officials: Suk Jin Kim, MD, PhD, Study Director — Samsung Medical Center, Seoul, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea